CLINICAL TRIAL: NCT07354334
Title: The Effect of Listening to Surah Al-Inshirah in the Early Postpartum Period After Cesarean Birth on Women's Spiritual Well-Being, Depression, and Maternal Attachment: A Randomized Controlled Trial
Brief Title: Effect of Listening to Surah Al-Inshirah After Cesarean Birth on Postpartum Outcomes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Yasemin ERKAL AKSOY, Assoc. Dr., Selcuk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 22051998
Record Dates: First submitted 2026-01-12; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Postpartum Depression; Maternal-Fetal Relations; Spirituality
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either an intervention group receiving routine postpartum care plus listening to Surah Al-Inshirah or a control group receiving routine postpartum care only.
Masking Description: This is an open-label study. Due to the nature of the audio-based spiritual intervention, participants and researchers are aware of group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Surah Al-Inshirah Listening Group (Experimental): Participants in this group will receive routine postpartum care and will additionally listen to an audio recording of Surah Al-Inshirah during the early postpartum period following cesarean birth.
  Interventions: Behavioral: Listening to Surah Al-Inshirah
- Control (No Intervention): Participants in this group will receive routine postpartum care only, without any additional audio or spiritual intervention.

INTERVENTIONS:
Behavioral: Listening to Surah Al-Inshirah — Participants will listen to a standardized audio recording of Surah Al-Inshirah in a quiet and comfortable environment during the first 48 hours after cesarean birth, in addition to routine postpartum care.
  Arms: Experimental: Surah Al-Inshirah Listening Group

SUMMARY:
This randomized controlled trial aims to evaluate the effect of listening to the recitation of Surah Al-Inshirah during the early postpartum period after cesarean birth on women's spiritual well-being, depression levels, and maternal attachment. The postpartum period is a sensitive phase characterized by physical recovery, emotional changes, and adaptation to the maternal role, particularly following cesarean delivery. Spiritual and religious practices are commonly used as coping strategies in this period, especially in Muslim populations.

In this study, women who have undergone cesarean birth will be randomly assigned to either an intervention group or a control group. The intervention group will listen to the recitation of Surah Al-Inshirah in addition to receiving routine postpartum care, while the control group will receive routine postpartum care only. Outcomes related to spiritual well-being, postpartum depression, and maternal attachment will be assessed within the first 48 hours after birth. The findings of this study are expected to contribute to evidence-based, culturally sensitive, and low-cost supportive care practices in the early postpartum period.

DETAILED DESCRIPTION:
The postpartum period is a critical transition phase in which women experience significant physiological, psychological, and emotional changes. Women who give birth by cesarean section may face additional challenges such as postoperative pain, limited mobility, delayed recovery, and increased vulnerability to emotional distress. These factors may negatively affect spiritual well-being, increase the risk of postpartum depression, and interfere with the development of maternal attachment.

Spiritual care interventions have gained increasing attention as supportive approaches in maternal health, particularly in cultures where religious beliefs and practices play an important role in coping with stress and emotional difficulties. In Islamic tradition, listening to the recitation of the Qur'an is believed to promote inner peace, emotional comfort, and spiritual strength. Surah Al-Inshirah, which emphasizes relief after hardship and emotional ease, may be especially meaningful during the early postpartum period.

This study is designed as a randomized controlled trial and will be conducted in the postpartum wards of a tertiary hospital. The study population will consist of primiparous women aged 18 years and older who have undergone cesarean birth and meet the inclusion criteria. Participants will be randomly assigned to either the intervention group or the control group using a randomization procedure conducted by an independent healthcare professional to minimize allocation bias.

Women in the intervention group will receive routine postpartum care and will additionally listen to a standardized audio recording of Surah Al-Inshirah during the first 48 hours after birth. The recitation will be delivered in a calm and comfortable environment at a safe sound level, with multiple listening sessions scheduled during the early postpartum period. Women in the control group will receive routine postpartum care only, without any additional audio or spiritual intervention.

Data will be collected using a personal information form and validated measurement tools, including the Spirituality Index of Well-Being, the Edinburgh Postpartum Depression Scale, and the Maternal Attachment Scale. Measurements will be conducted at baseline and repeated approximately 48 hours after birth to assess changes in outcomes. Statistical analyses will be performed to compare outcomes between the intervention and control groups.

This study aims to provide scientific evidence regarding the effectiveness of a culturally appropriate, low-cost, and non-invasive spiritual intervention to support women's psychological and emotional well-being after cesarean birth. The results may inform holistic and culturally sensitive postpartum care practices in maternal and newborn health services.

ELIGIBILITY:
Inclusion Criteria:

* Being literate
* Able to speak and understand Turkish
* Aged 18 years or older
* Primiparous women
* Having undergone cesarean birth
* Gestational age at birth between 37 and 42 weeks
* Identifying as Muslim
* Willing to participate voluntarily after providing written informed consent
* Women who have given birth within the last 48 hours and are hospitalized during the early postpartum period

Exclusion Criteria:

* Having a diagnosed psychiatric disorder
* Newborn admitted to the neonatal intensive care unit
* Experiencing stillbirth
* Having a hearing impairment

Criteria for Withdrawal From the Study

* Development of obstetric complications for any reason during the study
* Requesting to withdraw from the study during the data collection process
* Reporting feeling unwell or uncomfortable during the data collection process

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 172 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Postpartum Depression Level | Within the first 48 hours postpartum
  Postpartum depression will be assessed using the Edinburgh Postnatal Depression Scale (EPDS), a validated self-report questionnaire measuring depressive symptoms in the postpartum period. Higher scores indicate higher levels of depressive symptoms.

SECONDARY OUTCOMES:
Spiritual Well-Being | Within the first 48 hours postpartum
  Spiritual well-being will be measured using the Spirituality Index of Well-Being (SIWB), which assesses individuals' perceived spiritual quality of life and sense of meaning and peace.
Maternal Attachment | Within the first 48 hours postpartum
  Maternal attachment will be evaluated using the Maternal Attachment Scale, which measures the emotional bond between mother and infant.